CLINICAL TRIAL: NCT05860361
Title: Advanced Proton Therapy Approaches: a Multicenter High-quality Data Registry
Status: Recruiting | Type: Observational
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: R1760722-IEO 1885
Record Dates: First submitted 2023-04-07; First posted 2023-05-16 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2023-06

CONDITIONS: Cancer
Keywords: proton therapy; registry; high-quality dataset; prospective data collection; hypofractionation
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Blood and saliva samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the present registry is to prospectively collect data on patients treated with protontherapy in order to improve knowledge on indication, feasibility, and clinical results of hypofractionated schedules applied in the setting of patients.

DETAILED DESCRIPTION:
Paucity and low evidence level data on protontherapy (PT) represent one of the main issues for the establishment of solid indications in the PT setting. Aim of the present registry is to provide a tool for systematic, prospective, harmonized, and multidimensional high-quality data collection to promote knowledge in the field of PT with a particular focus on the use of hypofractionation.

All patients with any type of oncologic disease (benign and malignant disease) who will be eligible for PT at the European Institute of Oncology (IEO), will be included in the present registry. Three levels of data collection will be implemented: Level 1 clinical research (patients outcome and toxicity, quality of life, and cost/effectiveness analysis); Level 2 radiological research (radiomic and dosiomic analysis, as well as biological modeling); Level 3 Biological and Translational research (biological biomarkers and genomic data analysis).

Endpoints and outcome measures of hypofractionation schedules will be evaluated in terms of either Treatment Efficacy (tumor response rate, time to progression/percentages of survivors/median survival, clinical, biological, and radiological biomarkers changes, identified as surrogate endpoints of cancer survival/response to treatment) and Toxicity.

The study protocol has been approved by the IEO ethical committee (IEO 1885). Other than patients treated at IEO, additional PT facilities (equipped with IBA Proteus®ONE or Proteus®PLUS technologies) are planned to join the registry data collection. Moreover, the registry will be also fully integrated into international PT data collection networks.

ELIGIBILITY:
Inclusion criteria:

* diagnosis of oncological disease (benign and malignant disease);
* candidates to proton therapy;
* able to provide informed consent.

Exclusion criteria:

- age < 18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients aged >= 18 years with any type of oncologic disease (benign and malignant disease) eligible for proton therapy and able to provide informed consent (themselves, or through a designated legal guardian) to the registry.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2023-04-14 (Actual); Primary Completion 2028-10-01 (Estimated); Study Completion 2030-10-01 (Estimated)

PRIMARY OUTCOMES:
Treatment Efficacy: tumor response rate | 10 years
  tumor response rate according to RECIST criteria
Treatment Efficacy: % of tumor recurrence | 10 years
  % of tumor recurrence assessed by progression-free survival rate
Treatment Efficacy: rate of death | 10 years
  rate of death assessed by overall survival rates

SECONDARY OUTCOMES:
Treatment Toxicity: incidence of acute and late toxicity | 10 years
  incidence of acute and late toxicity collected according to CTCAE v. 6.0
Treatment Toxicity: patients quality of life | 10 years
  patients quality of life assessed by internationally validated EORTC questionnaires
Treatment Toxicity: patients pain | 10 years
  patients pain assessed by Visual Analog Score
Treatment Toxicity: treatment costs | 10 years
  treatment costs assessed with quality adjusted life years (QALY)

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Orecchia, Principal Investigator — European Institute of Oncology
Locations (1):
- European Institute of Oncology, Milan, Italy

IPD SHARING:
Plan to Share IPD: No